CLINICAL TRIAL: NCT04754490
Title: Exploring Patterns of Speech and Breathing to Indicate the Presence of Obstructive Disease
Brief Title: Exploring Breathing Patterns
Acronym: EPISODE
Status: Suspended | Type: Observational
Why Stopped: COVID 19
Sponsor: Cwm Taf University Health Board (NHS) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 256266
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Speech Recognition — Speech Recognition

SUMMARY:
Study Title Exploring patterns of speech and breathing to indicate the presence of obstructive respiratory disease.

Study Design Prospective Case Control Study Study Participants Participants will be patients attending the respiratory physiology clinic at the Cardiopulmonary Unit, Prince Charles Hospital for an assessment of their lung function. In addition a cohort of control participants without obstructive respiratory disease will be recruited with the assistance of the British Lung Foundation charity.

Planned Size of Sample (if applicable) We have received funding for 52 ½ day sessions and we plan to recruit on average 2 participants per session. As such we aim to recruit a minimum of 100 participants. In addition we are working with the British Lung Foundation to recruit a smaller Cohort of control participants and aim to recruit a minimum of 25 control participants.

Planned Study Period Jan 2019 - Aug 2019 Research Aim(s) This primary objective of this novel study it to create an anonymised database of speech patterns of patients with chronic respiratory disease and healthy aged matched controls for comparison with lung function and medical history.

The primary aims are to:

* Collect breathing patterns from individuals under a range of talking modalities
* Understand how easy it is to gather short speech recordings
* Explore the preferences of patients to be recorded talking

ELIGIBILITY:
6.1.2 Inclusion criteria Patient Participants

1. Adult patient >18 years old referred for spirometry in the Respiratory Physiology Clinic at Prince Charles Hospital;
2. Clinically defined obstructive or restrictive respiratory disease (indicated by spirometry)
3. Clinically stable (indicated by being able to undergo spirometry)
4. No significant unstable disease co-morbidities (indicated by being able to undergo spirometry)
5. Capable of providing informed consent.
6. Willing to take part in all study measurements.
7. The speaking exercise will be conducted in English on this study.
8. Participants are not taking part in any other research. 6.1.3 Inclusion criteria Control Participants

1. No obstructive or restrictive respiratory disease (indicated by spirometry) 2. Clinically stable (indicated by being able to undergo spirometry) 3. No significant unstable disease co-morbidity's (indicated by being able to undergo spirometry) 4. Capable of providing informed consent. 5. Willing to take part in all study measurements. 6. The speaking exercise will be conducted in English on this study. 7. Participants are not taking part in any other research.

6.1.4 Exclusion criteria for both Patient and Control Participants

1. Any form of challenge testing in the Respiratory Physiology Department involving salbutamol.
2. Severe Sensory and/or Cognitive Impairment
3. Inability to complete study measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patient >18 years old referred for spirometry in the Respiratory Physiology Clinic at Prince Charles Hospital;
  Eligibility Criteria - Control Participants Control participants will be contact through the British Lung Foundations local groups who have indicated their willingness to be involved in local clinical research to act as control participants. As all prospective participants will have had their respiratory function measured before taking part by a Respiratory Physiologist, we do not expect to have to screen for medical issues for participation in the study. Furthermore, the actual tests the participants will be undertaking will be non - invasive, submaximal and will require little or no effort.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Collect breathing patterns from individuals under a range of talking modalities | less than 5 minutes
  breathing pattern
Understand how easy it is to gather short speech recordings | 3 minutes
  verbal description
Explore the preferences of patients to be recorded talking | 3 minutes
  verbal description

CONTACTS AND LOCATIONS:
Locations (1):
- Cwm Taf Morgannwg Health Board, Abercynon, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No